CLINICAL TRIAL: NCT00320060
Title: A Randomized, Double-Blind, Placebo-Controlled, Multi-Center, 24-Week Study to Evaluate the Safety and Tolerability of Pyridorin (Pyridoxamine Dihydrochloride) in Patients With Diabetic Nephropathy Associated With Type 1 or Type 2 Diabetes
Brief Title: Effect of Pyridorin in Patients With Diabetic Nephropathy
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: BioStratum (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: PYR-206
Record Dates: First submitted 2006-04-27; First posted 2006-04-27 (Estimated); Last update posted 2006-04-27 (Estimated); Status verified 2006-04

CONDITIONS: Diabetic Nephropathy
Keywords: Diabetic nephropathy; Advanced Glycation Endproduct Inhibitor; Pyridorin; Pyridoxamine
MeSH Terms: conditions — Diabetic Nephropathies | interventions — pyridoxamine dihydrochloride

INTERVENTIONS:
Drug: Pyridorin (pyridoxamine dihydrochloride)

SUMMARY:
The primary objective of the study is to evaluate the safety and tolerability of Pyridorin (pyridoxamine dihydrochloride) 50 mg given orally twice daily in patients with diabetic kidney disease.

ELIGIBILITY:
Inclusion Criteria:

* Males and Females (non-pregnant and non-lactating) between 18 and 70 years of age with type 1 or type 2 diabetes
* Sitting blood pressure of <=170/100 mm Hg at weeks -2 and -1
* Hemoglobin A1C <=12% at week -2
* Patients with diagnosis of diabetic nephropathy as defined by

  1. Serum Creatinine <=2.0 mg/dL at weeks -2 and -1
  2. Urinary albumin excretion >=300 mg/24 hours at week -2
  3. Diagnosis of diabetic retinopathy
* Creatinine clearance >=40 mL/min at weeks -2 and -1
* Voluntary written consent to participate in this study

Exclusion Criteria:

* History of allergic or adverse response to any B vitamin
* History of major cardiovascular or cerebrovascular events
* History of cancer except adequately treated basal or squamous cell carcinoma of the skin
* History of diabetic ketoacidosis

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 128
Dates: Start 2001-10; Study Completion 2003-01

CONTACTS AND LOCATIONS:
Overall Officials: Thorsten P Degenhardt, Ph.D., Study Director — BioStratum, Inc.